CLINICAL TRIAL: NCT04696198
Title: Thoracic Mobility in Cystic Fibrosis Care
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Göteborg University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: FoU i VGR: 272 800
Record Dates: First submitted 2021-01-04; First posted 2021-01-06 (Actual); Last update posted 2024-02-29 (Actual); Status verified 2024-02

CONDITIONS: Cystic Fibrosis
Keywords: Rib cage; Range of motion; Pain; Spirometry
MeSH Terms: conditions — Cystic Fibrosis; Pain | interventions — Standard of Care

STUDY DESIGN:
Intervention Model Description: The patients are randomized to either of the groups, intervention or delayed intervention.
Who Masked: Outcomes Assessor
Masking Description: The outcome assessor will be blinded
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Range of motion (Experimental): Treatment is based on a set diagnostic and therapeutic protocol and carried out by registered health care professionals that are additionally trained in manual therapy intervention. 30 minutes of treatment will be given once a week over a period of two months
  Interventions: Other: Manual Therapy Intervention
- Standard care (Other): Standard care
  Interventions: Other: Standard care

INTERVENTIONS:
Other: Manual Therapy Intervention — Manual Therapy Interventions to improve range of motion and decrease pain
  Arms: Range of motion
Other: Standard care — standard care
  Arms: Standard care

SUMMARY:
Cystic fibrosis (CF) is an inherited, genetic disease of the body's mucus-producing glands that primarily affects the lungs and gastrointestinal tract. There are no studies that have examined anatomical changes, the connection between structure and function in the ribcage and the effect of symptom-relieving manual treatment.

The purpose of the study is therefore to investigate chest mobility in people with CF.

Method The study is conducted in three parts; a / A retrospective longitudinal part whose purpose is to investigate possible changes in the chest configuration in relation to deterioration of lung volumes in a cohort of CF patients. Chest configuration will be measured standardized and blinded on computed tomography (CT) images and related to results from spirometry examinations.

b / A prospective, consecutive cross-sectional study of the same cohort. The aim is to investigate the extent of stiffness and pain that is examined standardized (number of pain-free / normal moving structures) and its relation to objective examination of respiratory movements, respiratory muscle strength and spirometry.

c / A randomized controlled single-blind study aimed at evaluating the effect of manual treatment for pain and reduced mobility in patients with these symptoms. The treatments consist of standardized manual therapy with passive joint mobilization without impulse and soft tissue treatment. Evaluation will be done via the examination protocol in sub-study b / as well as objective measurements of respiratory movements (primary variable), respiratory muscle strength and spirometry which will be performed by a blinded tester both before and immediately after the intervention / control period.

Clinical significance When it comes to CF care, great medical advances have been made and for Swedish patients, the physiotherapeutic active treatment has proven to have very good effects. However, there are areas where care can be improved. The results from our study will provide additional breadth to strategies in CF care

ELIGIBILITY:
Inclusion Criteria:

* Diagnosed with cystic fibrosis
* >18 years of age

Exclusion Criteria:

* participation in clinical trials or other interventional studies, or, medical conditions that -as judged by the medical doctor in charge contraindicates the proposed intervention.

Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 63 (Actual)
Dates: Start 2019-09-09 (Actual); Primary Completion 2023-10-31 (Actual); Study Completion 2023-10-31 (Actual)

PRIMARY OUTCOMES:
Manual examination | Two months after inclusion
  Pain and stiffness in the ribcage according to a specific and tested form

SECONDARY OUTCOMES:
Vital capacity | Two months after inclusion
  Spirometry
Forced vital capacity during one second | Two months after inclusion
  Spirometry
Respiratory Muscle Strength | Two months after inclusion
  Maximum inspiratory and expiratory pressure
Respiratory movements | Two months after inclusion
  By Respiratory Movement Measuring Instrument
Patient Specific Functional Scale, PSFS | Two months after inclusion
  Function during individual activities. Ability to perform the individual activities are scored on a scale from 0 (not able to perform) to 10 (totally able to perform).

CONTACTS AND LOCATIONS:
Overall Officials: Monika Fagevik Olsén, PhD, Principal Investigator — Sahlgrenska University Hospital
Locations (1):
- Göteborg University, Gothenburg, Sweden

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Sinderholm Sposato N, Bjersa K, Gilljam M, Lannefors L, Fagevik Olsen M. Effectiveness of manual therapy interventions in cystic fibrosis care: a pilot study. J Bodyw Mov Ther. 2024 Jul;39:323-329. doi: 10.1016/j.jbmt.2024.02.036. Epub 2024 Mar 12. PMID 38876647